CLINICAL TRIAL: NCT03712059
Title: National Colorectal Polyp Care for Diagnosis, Classification and Resection
Brief Title: National Colorectal Polyp Care
Acronym: NCPC
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: 175 medical centers in China (Ambiguous)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept and Digestive Endoscopy Center, Changhai Hospital
Other Study IDs: NCPC
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Polyp
Keywords: Colorectal neoplasia; Polypectomy; Artificial intelligence
MeSH Terms: interventions — Colonoscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Screening group: All patients receive FIT test and colonoscopy, whose age, sex, family history, smoking history, body mass index (BMI), diabetes and other risk factors are collected by researchers through pad, equipped with a specially designed database and app. Using colonoscopy results as the gold standard, the diagnostic value of risk prediction model for the Chinese population is explored, and the optimal strategy of colonoscopy practice for the Chinese established initially.
  Interventions: Diagnostic Test: FIT test and colonoscopy
- Adenoma resection group: During the polypectomy of 2000 patients, for all pathologically confirmed or NBI-predicted adenomas with size<10mm, 1-2 biopsies were randomly performed on the edge after resection to determine the completion rate of the polypectomy.
  Interventions: Diagnostic Test: Polypectomy and biopsy
- Identification and classification group: For 12000 patients regardless of cancer diagnosis or polypectomy, if there is polyp, NBI (magnification) observation is required, with 4 white light and NBI images collected and reserved, respectively. If there is magnifying endoscopy, another 4 endoscopic images of magnification are also required. Endoscopists are invited to predict the pathology of polyps according to the NICE classification principle and endoscopic images, and upload the pathological results and endoscopic images within 2-4 week after colonoscopy.
  Interventions: Diagnostic Test: FIT test and colonoscopy; Diagnostic Test: Polypectomy and biopsy; Diagnostic Test: Classification

INTERVENTIONS:
Diagnostic Test: FIT test and colonoscopy — All included patients received FIT test and then colonoscopy, with the risk factors of CRC recorded. The diagnostic performance of predicting model (based on FIT and risk factors) and colonoscopy were compared.
  Groups: Identification and classification group; Screening group
Diagnostic Test: Polypectomy and biopsy — All included patients received polypectomy, and then biopsy is performed on the edge of resection for patients with < 10 mm adenoma (confirmed by pathology or predicted by NBI images), with the complete resection rate of polyps being calculated.
  Groups: Adenoma resection group; Identification and classification group
Diagnostic Test: Classification — Pathology of polyps is classified by endoscopists through NICE principle and the performance of classification between endoscopists and computer is compared.
  Groups: Identification and classification group

SUMMARY:
This study has three main purposes：screening: the first purpose is to evaluate the diagnostic value of combintion of the life risk factors and immunochemical fecal occult blood test (FIT) on detection of colorectal neoplasia in Chinese population; resection: the second objective is to investigate the complete resection rate of colorectal adenoma and risk factors of incomplete resection in China; identification and classification: the third objective is to initially establish an artificial intelegence-assissted recognition and classification system of polyp based on deep learning.

DETAILED DESCRIPTION:
This study is a multi-center cross-sectional survey and diagnostic test led by the National Clinical Research Center for Digestive Disease (Shanghai) (Department of Gastroenterology, Changhai Hospital, Naval Medical University), which is conducted at about 175 digestive endoscopy centers nationwide in China, with the expectation of including 12,000 patients (10,000 screenig and 2,000 adenoma resection). The basic characteristics of patients, bowel preparation method and quality, and related information of colonoscopy are recorded in detail. According to the research purpose, the whole project can be divided into three sections.

1. Screening section: All patients receive FIT test and colonoscopy, whose age, sex, family history, smoking history, body mass index (BMI), diabetes and other risk factors are collected by researchers through pad, equipped with a specially designed database and app. Using colonoscopy results as the gold standard, the risk prediction model for the Chinese population is explored, and the optimal strategy of colonoscopy practice for the Chinese established initially.
2. Resection section: During the polypectomy, for all pathologically confirmed or NBI-predicted adenomas with size<10mm, 1-2 biopsies were randomly performed on the edge after resection to determine the completion rate of the polypectomy.
3. Identification and classification section: For Patients regardless of cancer diagnosis or polypectomy, if there is polyp, observation of narrow band imaging (NBI) with or without magnification is required, with 4 white light and NBI images collected and reserved, respectively. If there is magnifying endoscopy, another 4 endoscopic images of magnification are also required. Endoscopists are invited to predict the pathology of polyps according to the NBI International Colorectal Endoscopic (NICE) classification principle and endoscopic images, and upload the pathological results and endoscopic images within 2-4 week after colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old and patients with or without alarming gastrointestinal symptoms were analyzed separately.
2. 3-4 L polyethylene glycol and foaming agent are used for bowel preparation.
3. Withdrawal time ≥6mins (excluding the time of biopsy)

Exclusion Criteria:

1. A history of acute myocardial infarction (within 6 months), severe heart, liver, kidney dysfunction, or mental illness.
2. Patients taking anticoagulants such as aspirin and warfarin, or who have coagulopathy.
3. Patients with inflammatory bowel disease and colon polyposis.
4. History of colonic procedure (including surgery, polypectomy, EMR, and ESD) in the screening section
5. Diameter of polyp greater than 1cm, lateral developmental lesions (LST), colon cancer, lesions requiring ESD and surgery
6. Patients participating in other clinical trials now or within 60 days.
7. Intestinal obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who referred to the outpatient and received colonoscopy.
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Detection of colorectal neoplasia | 24 hours
  Colorectal neoplasia included CRCs, adenomas, sessile serrated adenomas/polyps, traditional serrated adenomas/polyps, and hyperplastic polyps ≥10 mm, which were recommended to have a shorter surveillance interval after polypectomy

SECONDARY OUTCOMES:
Complete resection rate of polypectomy | 24 hours
Specificity and sensitivity of endoscopists and artificial intelligence-assisted system in classifying polyps | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yeoh KG, Ho KY, Chiu HM, Zhu F, Ching JY, Wu DC, Matsuda T, Byeon JS, Lee SK, Goh KL, Sollano J, Rerknimitr R, Leong R, Tsoi K, Lin JT, Sung JJ; Asia-Pacific Working Group on Colorectal Cancer. The Asia-Pacific Colorectal Screening score: a validated tool that stratifies risk for colorectal advanced neoplasia in asymptomatic Asian subjects. Gut. 2011 Sep;60(9):1236-41. doi: 10.1136/gut.2010.221168. Epub 2011 Mar 14. PMID 21402615
- [Background] Wong MC, Lam TY, Tsoi KK, Hirai HW, Chan VC, Ching JY, Chan FK, Sung JJ. A validated tool to predict colorectal neoplasia and inform screening choice for asymptomatic subjects. Gut. 2014 Jul;63(7):1130-6. doi: 10.1136/gutjnl-2013-305639. Epub 2013 Sep 17. PMID 24045331
- [Background] Sung JJ, Ng SC, Chan FK, Chiu HM, Kim HS, Matsuda T, Ng SS, Lau JY, Zheng S, Adler S, Reddy N, Yeoh KG, Tsoi KK, Ching JY, Kuipers EJ, Rabeneck L, Young GP, Steele RJ, Lieberman D, Goh KL; Asia Pacific Working Group. An updated Asia Pacific Consensus Recommendations on colorectal cancer screening. Gut. 2015 Jan;64(1):121-32. doi: 10.1136/gutjnl-2013-306503. Epub 2014 Mar 19. PMID 24647008
- [Background] Chiu HM, Ching JY, Wu KC, Rerknimitr R, Li J, Wu DC, Goh KL, Matsuda T, Kim HS, Leong R, Yeoh KG, Chong VH, Sollano JD, Ahmed F, Menon J, Sung JJ; Asia-Pacific Working Group on Colorectal Cancer. A Risk-Scoring System Combined With a Fecal Immunochemical Test Is Effective in Screening High-Risk Subjects for Early Colonoscopy to Detect Advanced Colorectal Neoplasms. Gastroenterology. 2016 Mar;150(3):617-625.e3. doi: 10.1053/j.gastro.2015.11.042. Epub 2015 Nov 25. PMID 26627608
- [Background] Pohl H. Polyp resection - lessons learned. Endoscopy. 2013 Dec;45(12):1030-1. doi: 10.1055/s-0033-1358830. Epub 2013 Nov 28. No abstract available. PMID 24288223
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Gupta N, Bansal A, Rao D, Early DS, Jonnalagadda S, Wani SB, Edmundowicz SA, Sharma P, Rastogi A. Prevalence of advanced histological features in diminutive and small colon polyps. Gastrointest Endosc. 2012 May;75(5):1022-30. doi: 10.1016/j.gie.2012.01.020. Epub 2012 Mar 9. PMID 22405698
- [Background] Hassan C, Pickhardt PJ, Kim DH, Di Giulio E, Zullo A, Laghi A, Repici A, Iafrate F, Osborn J, Annibale B. Systematic review: distribution of advanced neoplasia according to polyp size at screening colonoscopy. Aliment Pharmacol Ther. 2010 Jan 15;31(2):210-7. doi: 10.1111/j.1365-2036.2009.04160.x. Epub 2009 Oct 8. PMID 19814745
- [Background] Hassan C, Pickhardt PJ, Rex DK. A resect and discard strategy would improve cost-effectiveness of colorectal cancer screening. Clin Gastroenterol Hepatol. 2010 Oct;8(10):865-9, 869.e1-3. doi: 10.1016/j.cgh.2010.05.018. Epub 2010 Jun 1. PMID 20621680
- [Background] McGill SK, Evangelou E, Ioannidis JP, Soetikno RM, Kaltenbach T. Narrow band imaging to differentiate neoplastic and non-neoplastic colorectal polyps in real time: a meta-analysis of diagnostic operating characteristics. Gut. 2013 Dec;62(12):1704-13. doi: 10.1136/gutjnl-2012-303965. Epub 2013 Jan 7. PMID 23300139
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Background] Rees CJ, Rajasekhar PT, Wilson A, Close H, Rutter MD, Saunders BP, East JE, Maier R, Moorghen M, Muhammad U, Hancock H, Jayaprakash A, MacDonald C, Ramadas A, Dhar A, Mason JM. Narrow band imaging optical diagnosis of small colorectal polyps in routine clinical practice: the Detect Inspect Characterise Resect and Discard 2 (DISCARD 2) study. Gut. 2017 May;66(5):887-895. doi: 10.1136/gutjnl-2015-310584. Epub 2016 Apr 19. PMID 27196576
- [Background] Esteva A, Kuprel B, Novoa RA, Ko J, Swetter SM, Blau HM, Thrun S. Dermatologist-level classification of skin cancer with deep neural networks. Nature. 2017 Feb 2;542(7639):115-118. doi: 10.1038/nature21056. Epub 2017 Jan 25. PMID 28117445
- [Background] Gulshan V, Peng L, Coram M, Stumpe MC, Wu D, Narayanaswamy A, Venugopalan S, Widner K, Madams T, Cuadros J, Kim R, Raman R, Nelson PC, Mega JL, Webster DR. Development and Validation of a Deep Learning Algorithm for Detection of Diabetic Retinopathy in Retinal Fundus Photographs. JAMA. 2016 Dec 13;316(22):2402-2410. doi: 10.1001/jama.2016.17216. PMID 27898976
- [Background] Hayashi N, Tanaka S, Hewett DG, Kaltenbach TR, Sano Y, Ponchon T, Saunders BP, Rex DK, Soetikno RM. Endoscopic prediction of deep submucosal invasive carcinoma: validation of the narrow-band imaging international colorectal endoscopic (NICE) classification. Gastrointest Endosc. 2013 Oct;78(4):625-32. doi: 10.1016/j.gie.2013.04.185. Epub 2013 Jul 30. PMID 23910062